CLINICAL TRIAL: NCT06040580
Title: The Use of Resting State fMRI and CSD Tractography for Pre-operative Brain Mapping: a Cross-sectional Study
Brief Title: Can we Use Resting-state fMRI and CSD Fiber Tractography for Presurgical Mapping?
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof dr Stefan Sunaert, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S61759
Record Dates: First submitted 2023-06-04; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Brain Tumor; Brain Pathology; Epilepsy; Vascular Malformations, Brain
Keywords: Functional MRI; Diffusion MRI; Fiber Tractography; Preoperative brain mapping
MeSH Terms: conditions — Brain Neoplasms; Epilepsy; Central Nervous System Vascular Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Preoperative patients in need of brain surgery for varying brain pathology who require presurgical brain mapping with MRI (fMRI, and dMRI)

SUMMARY:
This prospective study aims to investigate and validate the use of resting-state functional MRI (rs-fMRI) and high angular resolution diffusion imaging (HARDI), specifically constrained spherical deconvolution (CSD) tractography, for functional and structural brain mapping prior to neurosurgery. The goal is to assess the feasibility of replacing task-based fMRI (tb-fMRI) and diffusion tensor imaging (DTI) with fiber tractography (FT) using the fiber assignment by continuous tracking (FACT) algorithm. The study focuses on mapping sensory-motor, language, visual, and higher cognitive functional and structural networks in patients with brain pathology suitable for surgical intervention. The objective is to improve neurosurgical planning, navigation, and risk assessment through the utilization of rs-fMRI and CSD tractography.

DETAILED DESCRIPTION:
This study aims to prospectively investigate and validate the application of resting state functional MRI (rs-fMRI) and High angular resolution diffusion imaging (HARDI), particularly constrained spherical deconvolution (CSD) tractography, in presurgical functional and structural brain mapping for the purposes of neurosurgical planning, navigation and risk assessment. The main objective is to determine whether rs-fMRI and CSD tractography are capable of replacing task based fMRI (tb-fMRI) and diffusion tensor imaging (DTI) based fiber tractography (FT) using the fiber assignment by continuous tracking (FACT) algorithm for mapping the sensory-motor, language, visual, as well as higher cognitive functional and structural networks of the brain in patients with brain pathology amenable for surgical intervention. This research question will be investigated by acquiring tb-fMRI and rs-fMRI, as well as HARDI data for presurgical patients. The routine workflow of presurgical planning and risk assessment using tb-fMRI and DTI FT will be followed and used for the initial planning. Previous studies have revealed a high degree of concordance between rs-fMRI and tb-fMRI[1]-[5] as well as between CSD and DTI FT[6]-[8], but drew such conclusions from relatively small sample sizes. The aim is to incorporate the rs-fMRI and CSD results into the presurgical planning process albeit with more weight assigned to the tb-fMRI and DTI results. The study population will consist of 10 normal controls for MR imaging optimization purposes only, 150 presurgical patients from the UZ Leuven imaging department regardless of the exact type of pathology (space occupying lesions, epilepsy, vascular malformations etc.).

As tb-fMRI has previously been validated versus the gold standard of functional mapping, electrical cortical stimulation (ECS), while rs-fMRI has previously been validated against tb-fMRI. The same has been done comparing DTI and CSD. To our knowledge however, a comparative study with such a large and diverse study population attempting to cross validate all these modalities against the gold standard has not yet been done.

Image acquisition acceleration methods, such as parallel imaging (PI), simultaneous multislice acquisitions (SMS) and compressed sensing (CS) will be used whenever feasible. These acceleration methods can potentially be exploited to improve fMRI, and dMRI data quality as well as shorten acquisition time. In the case of fMRI, PI and SMS can be used to increase temporal resolution, temporal signal to noise ratio and even spatial resolution. dMRI stands to benefit from such techniques by increasing directional and/or spatial resolution.

ELIGIBILITY:
Inclusion Criteria:

* Stable clinical condition
* Cooperative and able to perform the fMRI tasks in question
* In need of preoperative MRI mapping scans

Exclusion Criteria:

* Absolute contraindications to MRI
* Previously underwent resective brain surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with any brain pathology amenable to surgery who have not undergone previous resective surgery, regardless of age, gender or type of disease.
  Healthy volunteers are only included for scan optimization puproses.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in accuracy between CSD and DTI fiber tractography as well as resting-state and task-based fMRI | Through phase 1 recruitment completion (about 2 years from start of recruitment)
  A comparative analysis examining differences in accuracy measures between different fMRI and dMRI tractography methods, namely resting-state fMRI v. task-based fMRI and DTI v CSD diffusion tractography using intraoperative direct electrical stimulation results as the ground truth

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No
Anonymized and coded data may be shared with other research groups upon reasonable request to the authors.

REFERENCES:
- [Background] Radwan AM, Sunaert S, Schilling K, Descoteaux M, Landman BA, Vandenbulcke M, Theys T, Dupont P, Emsell L. An atlas of white matter anatomy, its variability, and reproducibility based on constrained spherical deconvolution of diffusion MRI. Neuroimage. 2022 Jul 1;254:119029. doi: 10.1016/j.neuroimage.2022.119029. Epub 2022 Feb 26. PMID 35231632
- [Result] Radwan AM, Emsell L, Blommaert J, Zhylka A, Kovacs S, Theys T, Sollmann N, Dupont P, Sunaert S. Virtual brain grafting: Enabling whole brain parcellation in the presence of large lesions. Neuroimage. 2021 Apr 1;229:117731. doi: 10.1016/j.neuroimage.2021.117731. Epub 2021 Jan 14. PMID 33454411